CLINICAL TRIAL: NCT04254003
Title: Clinical Performance Evaluation of Two Daily Disposable Silicone Hydrogel Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: CLO870-C003
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Refractive Errors
Keywords: toric contact lens; daily disposable; silicone hydrogel contact lens; axis orientation; astigmatism
MeSH Terms: conditions — Refractive Errors; Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Test, then Control (Other): DT1 Toric contact lenses worn first, followed by AO1DfA contact lenses, as randomized. Each product will be worn in both eyes for approximately 1 hour.
  Interventions: Device: DT1 Toric contact lenses; Device: AO1DfA contact lenses
- Control, then Test (Other): AO1DfA contact lenses worn first, followed by DT1 Toric contact lenses, as randomized. Each product will be worn in both eyes for approximately 1 hour.
  Interventions: Device: DT1 Toric contact lenses; Device: AO1DfA contact lenses

INTERVENTIONS:
Device: DT1 Toric contact lenses — Delefilcon A contact lenses for the optical correction of astigmatism in people with healthy eyes with or without refractive ametropia (myopia or hyperopia)
  Other Names: Test; DAILIES TOTAL1 for Astigmatism (DT1 Toric)
Device: AO1DfA contact lenses — Senofilcon A contact lenses for the optical correction of astigmatism in people with healthy eyes with or without refractive ametropia (myopia or hyperopia)
  Other Names: Control; Acuvue Oasys 1-Day for Astigmatism (AO1DfA)

SUMMARY:
The purpose of this study is to evaluate the rotational behavior of DT1 Toric contact lenses.

DETAILED DESCRIPTION:
This is a single visit, non-dispense study where subjects will be exposed to the test and control lenses for approximately 1 hour each.

ELIGIBILITY:
Inclusion Criteria:

* Current wearer of any commercial soft daily wear contact lens with at least 3 months of wearing experience with a minimum wearing time of 5 days per week and 8 hours per day.
* Requiring contact lens (manifest refraction) of a cylindrical power of -0.75 to -2.50 diopter cylinder (DC).
* Best corrected distance visual acuity 20/25 or better Snellen in each eye (as determined by manifest refraction at screening).
* Willing to NOT use rewetting/lubricating drops at any time during the study. Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any anterior segment infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the Investigator.
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the Investigator.
* History of refractive surgery or plan to have refractive surgery during the study or irregular cornea in either eye.
* Eye injury in either eye within 12 weeks immediately prior to enrollment for this trial.

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Percent of DT1 toric lenses with axis orientation within ±30° from the intended axis, 10 min after lens insertion | Day 1, 10 minutes after lens insertion, each product
  A slit lamp will be used to observe axis orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (2):
- United States (2):
  - Alcon Investigative Site CT-11, Maitland, Florida
  - Alcon Investigative Site CT-27, Eden Prairie, Minnesota

IPD SHARING:
Plan to Share IPD: No